CLINICAL TRIAL: NCT05445635
Title: Added Value of a Small Camera (Iriscope) in the Endoscopic Diagnosis of Peripheral Lung Nodules and Masses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Taton, Doctor, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P2021/770
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Nodule, Solitary
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iriscope (Experimental)
  Interventions: Device: Iriscope
- EBUS (Active Comparator)
  Interventions: Device: Iriscope
- Combined Iriscope + EBUS (Experimental)
  Interventions: Device: Iriscope

INTERVENTIONS:
Device: Iriscope — The use of Iriscope to improve the diagnostic yield of bronchoscopy in the setting of peripheral lung nodules

SUMMARY:
Since the beginning of lung screening program in the different countries around the world by chest CT scan, numerous lung nodules and masses of unknown etiology are diagnosed.

Usually, the pathological diagnosis is obtained by bronchoscopy. However, peripheral bronchi cannot be seen after the fifth bronchial division as the diameter of the broncoscope is greated than the diameter of the bronchi. Therefore, the Iriscope was developed. It consists in a thin catheter with a mini-camera at its distal extremity.

The aime of this study is to evaluate the diagnostic yield of bronchoscopy guided by Iriscope in the setting of peripheral lung nodules and masses supect of malignancy, to compare the Iriscope to endobronchial radial ultrasonography (which is a validated technique to guide bronchoscopy in the setting of peripheral lung nodules and masses) and to evaluate the added value on the diagnostic yield by combining these 2 techniques.

ELIGIBILITY:
Inclusion Criteria:

* Lung nodules or masses suspect of malignancy with a diameter between 2 and 5 centimeters

Exclusion Criteria:

* Any contraindication to general anesthesia
* Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of bronchoscopy | Pathological diagnosis just after the bronchoscopy. In case of unspecified diagnosis after bronchoscopy, a follow up may be performed by chest ct scan up to 6 months.
  The diagnosis will be obtained by pathological analysis. The diagnostic yield is the number of cases with a pathological diagnosis obtained by bronchoscopy on the total number of cases. In case of unspecified diagnosis, the fianal diagnosis will be given by the pathological naalysis of the surgical resection or chest CT follow up.

SECONDARY OUTCOMES:
Complications of bronchoscopy | Just after the bronchoscopy to 1 month after the procedure
  Number of participants that present a pneumothorax or hemorrhage after the bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Taton, Resident, Principal Investigator — Hôpital Erasme, Université Libre de Brussels, Brussels, Belgium
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided